CLINICAL TRIAL: NCT05948696
Title: To Explore the Experience of Patients With Chronic Schizophrenia Participating in Horticultural Group Therapy
Brief Title: Experience of Horticultural Group Therapy Among People With Chronic Schizophrenia
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: TsaoTun Psychiatric Center, Department of Health, Taiwan (Other)
Responsible Party: Principal Investigator, Ying-Jyun Shih, MSc, TsaoTun Psychiatric Center, Department of Health, Taiwan
Other Study IDs: AF007
Record Dates: First submitted 2023-07-08; First posted 2023-07-17 (Actual); Last update posted 2023-07-17 (Actual); Status verified 2023-07

CONDITIONS: Chronic Schizophrenia
Keywords: chronic schizophrenia, horticultural therapy group

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Horticultural participants: Inpatients with chronic schizophrenia who attend to a horticultural group therapeutic program.
  Interventions: Behavioral: Horticultural group therapy.

INTERVENTIONS:
Behavioral: Horticultural group therapy. — Estimated 10 persons with schizophrenia who attend to a 12-week horticultural group therapy will be assessed for their experience about the program.

SUMMARY:
Taiwan National Health Insurance Administration database shows that the number of people seeking medical treatment due to mental illness has reached 1.454 million in 2021. The annual growth rate of mental illness is between 3.3% to 6.6%. Fifty percent of mental illness patient has catastrophic illness certificate because of chronic schizophrenia (Ministry of Health and Welfare,2022). Auditory hallucinations, delusions, emotional disturbances, and disorder in behavior and the poor ability of speaking are common in patients with schizophrenia. These symptoms lead to reduce the cognitive and executive function, resulting severe impairment of eventual daily living functions and social interactions. Thus, the cost of hospitalization and medical fee is increased. It is worth considering the appropriateness of the model of care. According to researches, people with schizophrenia still strive to pursue a happy and satisfying life. However, statistics of satisfaction and happiness are still lower than people who are healthy (Palmer et al., 2014; Fervaha et al., 2016).

The American Horticultural Therapy Association (AHTA) pointed out that horticultural therapy increases the well-being of participants through active or passive participation in plant-related activities. It also helps participants learn new skills or regain lost skills. Furthermore, psychiatric symptoms, recovery outcomes, life satisfaction, and the benefits of social function are significantly improved (Lu et al., 2021; Oh et al., 2018). Taiwanese scholars mention that combining horticultural activities and group psychotherapy improves the therapeutic results. It means that using of flowers and plants in gardening combines with the therapeutic advantages of group psychotherapy, mental illness patients can benefit more from it (Lin, 2016).

This study aims to explore the experience of patients with chronic schizophrenia participating in horticultural group therapy. This research design adopts the purposive sampling in qualitative method from a psychiatric hospital in central Taiwan. It is expected that 10 participants will involve in 12 times of horticultural therapy, and recordings will be made in each group. After 12 times of the therapy, participants will be involved in semi-structured audio-recorded interviews. The collected data were analyzed step by step using the content analysis method. In addition, participants will finish the questionnaires of the "Mental Well-Being Scale"," Satisfaction With Life Scale ", " activity of daily living Scale ", Instrumental Activities of Daily Living Scale", and "Group Efficacy Observation Form" before and after the therapies. The data will be conducted with descriptive statistics, Pearson's correlation coefficient, Chi-square Test, Paired Sample t test by using SPSS 21.0 statistical software. This research hopes to understand the impact of horticultural treatments in people who suffer from chronic schizophrenia, and provides a reference to clinical teams.

ELIGIBILITY:
Inclusion Criteria:

* Persons with schizophrenia and have been hospitalized to for more than 6 months.
* Intact or minimal cognitive performance on SPMSQ.
* Mild to moderate severity on Brief Psychiatric Rating Scale.
* ADL score>65 on Barthel Index
* Moderate or low on the Warwick-Edinburg Mental Well-being scale

Exclusion Criteria:

* Those who are not able to comply with the requirements of the study

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Persons with schizophrenia and have been hospitalized to for more than 6 months.
Sampling Method: Non-Probability Sample
Enrollment: 10 (Estimated)
Dates: Start 2023-06-06 (Actual); Primary Completion 2023-09-06 (Estimated); Study Completion 2023-09-29 (Estimated)

PRIMARY OUTCOMES:
Well-being | 12 weeks
  Measured with the Warwick-Edinburg Mental Well-being scale

SECONDARY OUTCOMES:
Basic and instrumental activities of daily living | 12 weeks

OTHER OUTCOMES:
Group Efficacy | 12 weeks
  Measured by Group Efficacy Observation Form

CONTACTS AND LOCATIONS:
Locations (1):
- TsaoTun Psychiatric Center, Nantou City, Taiwan